CLINICAL TRIAL: NCT02588677
Title: Multicenter, Randomised, Double-blind, Placebo-controlled, Parallel Group, Phase 2/3 Study to Compare the Efficacy and Safety of Masitinib
Brief Title: Masitinib in Combination With Riluzole for the Treatment of Patients Suffering From Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AB Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AB10015
Record Dates: First submitted 2015-10-20; First posted 2015-10-28 (Estimated); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: Amyotrophic Lateral Sclerosis (ALS) - masitinib
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — masitinib; Riluzole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Masitinib (3.0) & Riluzole (Experimental): masitinib 3 mg/kg/day + riluzole
  Interventions: Drug: Riluzole; Drug: Masitinib (3.0)
- Masitinib (4.5) & Riluzole (Experimental): masitinib 4.5 mg/kg/day (2) + riluzole
  Interventions: Drug: Masitinib (4.5); Drug: Riluzole
- Placebo & Riluzole (Placebo Comparator): Matched placebo
  Interventions: Drug: Riluzole; Drug: Placebo

INTERVENTIONS:
Drug: Masitinib (4.5) — 4.5 mg/kg/day
  Other Names: AB1010
  Arms: Masitinib (4.5) & Riluzole
Drug: Riluzole
  Other Names: Rilutek
Drug: Placebo
  Other Names: Placebo Oral Tablet
  Arms: Placebo & Riluzole
Drug: Masitinib (3.0) — 3 mg/kg/day
  Other Names: AB1010
  Arms: Masitinib (3.0) & Riluzole

SUMMARY:
The objective is to compare the efficacy and safety of masitinib in combination with riluzole in the treatment of patients suffering from Amyotrophic Lateral Sclerosis (ALS).

DETAILED DESCRIPTION:
Masitinib is novel tyrosine kinase inhibitor that targets microglia and mast cells through inhibiting a limited number of kinases. Masitinib blocks microglia proliferation and activation, and mast cell-mediated degranulation, the release of cytotoxic substances that might further damage the motor nerves.

There are two distinct populations of ALS patients: population of "Normal progressors" and population of "Faster progressors". Targeted population for primary analysis is population of "Normal progressors".

"Normal progressors" are ALS patients whose progression of ALSFRS-R score before randomization is less than 1.1 point per month.

ELIGIBILITY:
Inclusion Criteria:

Main inclusion criteria:

1. Familial or sporadic ALS
2. Patient diagnosed with probable of definite ALS
3. Patient treated with a stable dose of riluzole (100 mg/day) for at least 30 days prior to screening

Exclusion Criteria:

1. Patient who underwent tracheostomy and/or gastrostomy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Actual)
Dates: Start 2013-04; Primary Completion 2016-12-05 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Change in Amyotrophic Lateral Sclerosis functional rating scale (ALSFRS)-Revised | From baseline to week 48
  The amyotrophic lateral sclerosis functional rating scale (ALSFRS), which is a Validated instrument that assesses the functional status and the disease progression in patients with amyotrophic lateral sclerosis (ALS)

SECONDARY OUTCOMES:
Change of Forced Vital Capacity (FVC) | From baseline to week 48
  Forced vital capacity (FVC) measures the volume of air expelled from the lungs during a quick, forceful breath.
Progression Free Survival | Time from the randomization date until the earliest date for a decline of more than 9-points in ALSFRS-R score, asssesd over a maximum of 60 months
  Progression Free Survival is defined as the time from the randomization date until the earliest date for a decline of more than 9-points in ALSFRS-R score
Overall Survival | Time from the randomization date until death, asssesd over a maximum of 60 months
  Overall survival is defined as time in months from the randomization date to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jesus S Mora, MD, Principal Investigator — Unidad de ELA, Hospital San Rafael, c/ Serrano, 199, 28016 Madrid, Spain
Locations (1):
- Hospital Carlos III, Madrid, Spain

REFERENCES:
- [Derived] Mora JS, Bradley WG, Chaverri D, Hernandez-Barral M, Mascias J, Gamez J, Gargiulo-Monachelli GM, Moussy A, Mansfield CD, Hermine O, Ludolph AC. Long-term survival analysis of masitinib in amyotrophic lateral sclerosis. Ther Adv Neurol Disord. 2021 Jul 19;14:17562864211030365. doi: 10.1177/17562864211030365. eCollection 2021. PMID 34457038